CLINICAL TRIAL: NCT04528394
Title: A Randomized Phase II Trial Evaluating Toxicity and Efficacy Between Proton and Photon for Nasopharyngeal Carcinoma
Brief Title: Proton Versus Photon Radiotherapy for Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Jiade J. Lu, Executive Vice-President, Shanghai Proton and Heavy Ion Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-HNCNS-2019-32
Record Dates: First submitted 2020-08-24; First posted 2020-08-27 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Intensity-modulated radiation therapy; Proton beam therapy; Carbon-ion radiotherapy; Toxicity; Survival; Disease control
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Photons; Protons

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Photon combined with Carbon ion (Experimental): The participants received photon: 56 Gy/28 Fx for high-risk area(CTVhigh), 50.4 Gy/28 Fx for lower neck low-risk area(CTVlow), plus carbon ion: 15-17.5 GyE/5 Fx for boost for visible tumors.
  Interventions: Radiation: Photon; Radiation: Carbon ion
- Proton combined with Carbon ion (Experimental): The participants received proton: 56 GyE/28 Fx for high-risk area(CTVhigh), 50.4 GyE/28 Fx for lower neck low-risk area(CTVlow), plus carbon ion: 15-17.5 GyE/5 Fx for boost for visible tumors.
  Interventions: Radiation: Proton; Radiation: Carbon ion

INTERVENTIONS:
Radiation: Photon — Photon combined with Carbon ion in Arm 1
  Arms: Photon combined with Carbon ion
Radiation: Proton — Proton combined with Carbon ion in Arm 2
  Arms: Proton combined with Carbon ion
Radiation: Carbon ion — Same dose and fractionation will be used in both arms.

SUMMARY:
The purpose of this study is to compare the toxicity and therapeutic efficacy of proton or photon combined with carbon ion radiotherapy for newly diagnosed nasopharyngeal carcinoma.Participants will be randomized to 2 arms. Arm 1, participants received photon combined with carbon ion radiotherapy group, Arm 2, participants received proton combined with carbon ion radiotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to compare the toxicity and therapeutic efficacy of photon or proton combined with carbon ion radiotherapy for newly diagnosed nasopharyngeal carcinoma.Participants will be randomized to 2 arms. Arm 1 participants received photon combined with carbon ion radiotherapy (photon: 56 Gy/28 Fx, plus carbon: 15-17.5 gray equivalent [GyE]/5 Fx for boost). Arm 2, participants received proton combined with carbon ion radiotherapy (proton: 56 GyE/28 Fx, plus carbon: 15-17.5 GyE/5 Fx for boost). Adverse events will be documented according to CTCAE v4.03.The response of treatment will be evaluated according to RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed Nasopharyngeal carcinoma(WHO II/III type).
* Age ≥ 18 and ≤ 70 years of age.
* Eastern Cooperative Oncology Group score: 0-1.
* Adequate laboratory values within 30 dyas of enrollment to study defined as follows: 1) neutrophil > 2000/mm^3; 2) platelet > 100,000/mm^3; 3) total bilirubin < 1.5mg/dl; 4) alanine aminotransferase/aspartate aminotransferase < 1.5 upper limit of normal; 5) SCr < 1.5mg/dl; creatinine clearance rate > 60ml/min.
* Willing to accept adequate contraception for women with childbearing potential.
* Willing to sign the written informed consent; Informed consent must be signed before the enrollment in the trial.

Exclusion Criteria:

* Presence of distant metastasis.
* Received radiotherapy for head and neck before.
* Received surgery(except for biopsy) for primary lesion or cervical lymph node.
* Previous history of malignant tumor (within 5 years) or simultaneous existence of multiple primary tumors.
* Presence of diseases (such as Sjögren syndrome) that may interfere evaluation of xerostomia.
* Accompanied with severe major organ dysfunction.
* Presence of mental disease that may influence the understanding of informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2019-04-29 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related Xerostomia (≥Grade 2) as assessed by NCI CTCAE v4.03 | Xerostomia (≥Grade 2) occurred at 6 months after completion of radiotherapy
  CTCAE refers to Common Terminology Criteria for Adverse Events, which is one of the most frequently used criteria for toxicity grading after anti-cancer treatment.

SECONDARY OUTCOMES:
Overall survival of all patients | From randomization to death, a median of 3 years.
Progression-free survival of all patients | From randomization to death or disease progression, a median of 3 years.
Local control | From randomization to local failure, a median of 3 years.
Regional control | From randomization to regional failure, a median of 3 years.
Distant control | From randomization to distant failure, a median of 3 year.
Treatment-related adverse events as assessed by NCI CTCAE v4.03 | Time interval from start to 3 months after completion of radiotherapy.
  Acute and late toxicities induced by radiation therapy other than xerostomia.

CONTACTS AND LOCATIONS:
Overall Officials: Jiade Lu, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center,Shanghai, SPHIC
Locations (1):
- Shanghai Proton and Heavy Ion Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data including baseline characteristics, treatment information and follow-up data on toxicity, survival and disease control will be shared.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within 5 years after the publication of the study
Access Criteria: Data may be shared with radiation oncologists who are interested in examining the efficacy and toxicity of nasopharyngeal carcinoma patients treated with particle beam radiotherapy. Pooled analysis comparing IMRT and particle beam radiotherapy will be of particular interest. Detailed study protocol should be emailed along with the request of the data. We may carefully review the study protocol, and data will only be shared with well-designed studies.